CLINICAL TRIAL: NCT05769179
Title: Comparison of Different Manual Therapy Approaches in Patients With Chronic Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, seyda toprak celenay, associate professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/03/03
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Massage group (Experimental): Massage group will be applied classic massage+cervical stabilisation exercises
  Interventions: Other: Massage group
- Connective tissue massage group (Experimental): Connective tissue group will be applied connective tissue massage+cervical stabilisation exercises
  Interventions: Other: Connective tissue massage group
- Mobilization group (Experimental): Mobilization group will be applied cervical mobilization techniques+cervical stabilisation exercises
  Interventions: Other: Mobilization group

INTERVENTIONS:
Other: Massage group — Massage group will be applied classic massage and cervical stabilisation exercises 3 days a week for 4 weeks
  Arms: Massage group
Other: Connective tissue massage group — Connective tissue massage group will be applied connective tissue massage and cervical stabilisation exercises 3 days a week for 4 weeks
  Arms: Connective tissue massage group
Other: Mobilization group — Mobilization group will be applied cervical mobilization techniques and cervical stabilisation exercises 3 days a week for 4 weeks
  Arms: Mobilization group

SUMMARY:
The aim of the study was to compare the effects of different manual therapy approaches on pain, cervical range of motion, balance, functional status and life quality in patients with chronic neck pain.

DETAILED DESCRIPTION:
Various physiotherapy and rehabilitation methods are applied in the treatment of patients with chronic neck pain. Clinical practice guidelines for individuals with chronic neck pain recommend both manual therapy and exercise therapy among conservative treatments. Manual therapy are methods that can be safely applied to soft tissues and joints. Both manual therapy and exercise applications have been shown to have positive effects on neck pain and function. Some studies in the literature have also shown that manual therapy methods have positive effects on balance. However, no study examining the effects of different manual therapy (classical massage, connective tissue massage, manual joint techniques) approaches applied to individuals with chronic neck pain on pain, cervical range of motion, balance, functional status and quality of life was found in the literature.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18-65.
* To participate in the study voluntarily.
* Having a complaint of neck pain for at least 3 months.

Exclusion Criteria:

* To have undergone cervical spine surgery
* Having cervical fracture and/or joint subluxation/dislocation
* Severe degenerative arthritis
* Having a neurological disease (Parkinson's disease, poliomyelitis, etc.) or an -inflammatory rheumatic disease (ankylosing spondylitis, rheumatoid arthritis, etc.)
* Presence of malignancy
* Having cord compression and signs
* Severe radiculopathy or myelopathy
* Positive vertebrobasilar artery test,
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-30 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | change from baseline at 4 weeks
  Pain intensity will be assessed with the Visual Analogue Scale (a 100 mm long horizontal line). Patient will be asked to score the pain he/she feels out of 10. The beginning of the figure is "0 "no pain", ending in "10 "there is unbearable pain".

SECONDARY OUTCOMES:
Pressure Pain Threshold | change from baseline at 4 weeks
  Pressure Pain Threshold will be assessed with a digital algometer device. The device that objectively measures the pain threshold will be used for the evaluation. The probe of the device will be pressed on the trapezius muscle. The first pain threshold felt will be recorded.
Cervical Range of Motion | change from baseline at 4 weeks
  Cervical range of motion will be evaluated with a goniometer in the sitting position. Neck flexion, extension, right-left lateral flexion and right-left rotation ranges of motion will be recorded
Balance | change from baseline at 4 weeks
  Balance will be evaluated with the Biodex Balance System Device. The individual is placed on a platform of the device that evaluates the ability to keep the centre of gravity on the support surface. Changes in the centre of gravity of the individual standing on this platform will be recorded with this device in static and dynamic, with eyes open and closed.
Functional Status | change from baseline at 4 weeks
  Functional Status will be assessed with Neck Disability Index. This index consists of 10 items. Each item was scored from 0 (no disability) to 5 (complete disability). The total score ranged from 0 (no disability) to 50 (total disability). As the score increased, disability increased and as the score decreased, disability decreased.
Life quality | change from baseline at 4 weeks
  Life quality will be assessed with Short Form-36 questionnaire. The questionnaire consists of 36 items. Scoring is done over 100 points and the scores are between 0 and 100 points for each sub-parameter. "0" is calculated as the worst value and "100" as the best value.

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Toprak Celenay, Principal Investigator — Ankara Yildirim Beyazıt University